CLINICAL TRIAL: NCT01250873
Title: LY2216684 and Sertraline Pharmacokinetic Interaction Study in Healthy Subjects
Brief Title: A Pharmacokinetic Study of the Coadministration of LY2216684 With Sertraline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12611; H9P-EW-LNCT (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2216684/sertraline/LY2216684 + sertraline (Experimental): Period 1: LY2216684 18 milligram (mg) oral (po) dose on Days 1-3.
  Period 2: Sertraline 50 mg po dose on Day 4 followed by sertraline 100 mg po dose on Days 5-10.
  Period 3: LY2216684 18 mg po dose + sertraline 100 mg po dose on Days 11-13.
  Interventions: Drug: LY2216684; Drug: Sertraline

INTERVENTIONS:
Drug: LY2216684 — po administration
Drug: Sertraline — po administration

SUMMARY:
LY2216684 is being studied as adjunctive treatment for major depressive disorder (MDD) in participants who are partial responders to selective serotonin reuptake inhibitors (SSRIs). Sertraline is a medication that is widely used to treat MDD and is a known substrate of cytochrome P450s (CYP450s), including CYP450 2D6 (CYP2D6), CYP450 2C19 (CYP2C19), CYPP450 3A4 (CYP3A4), and a modest inhibitor of CYP2D6. Based on the diversity of hepatic metabolic clearance pathways for LY2216684 and its elimination by the kidney, it is expected that CYP2D6 inhibition by sertraline will not result in a substantial change in the pharmacokinetic (PK) profile of LY2216684. LY2216684 is only known to be a moderate inhibitor of CYP2C19, so it is unlikely that coadministration of sertraline with LY2216684 will result in a clinically meaningful change in the PK of sertraline. This study is being conducted to test these hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical history and physical examination.
* Male participants - Agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug.
* Female participants - Are women of child-bearing potential who test negative for pregnancy at the time of enrollment, have used a reliable method of birth control for 6 weeks prior to administration of study drug, and agree to use a reliable method of birth control during the study + 1 month following the last dose of study drug; or are women not of child-bearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause (at least 1 year without menses or 6 months without menses and a follicle stimulating hormone (FSH) level ≥40 mass International Units per milliliter (mIU/mL).
* Body mass index (BMI) up to 32.0 kilograms per square meter (kg/m^2).
* Have screening clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling according to the protocol.
* Have normal blood pressure and pulse rate (supine position and standing) as determined by the investigator.
* Are reliable and willing to be available for the duration of the study and willing to follow study procedures.
* Provided written informed consent approved by Lilly and the institutional review board (IRB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device, or off-label use of a drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies/intolerance to LY2216684, sertraline, or related compounds.
* Are persons who previously completed or discontinued from this study, or any other study investigating LY2216684 within 6 months prior to screening.
* Have a clinically significant abnormality in the 12-lead electrocardiogram (ECG) as determined by the investigator.
* Have significant history of or current cardiovascular (including dysrhythmias), respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have a history of seizure disorders.
* Have a history or presence of the signs and/or symptoms of hyponatremia.
* Have a history or presence of the signs and/or symptoms of hyperthyroidism as determined by an abnormal thyroid stimulating hormone (TSH) at screening.
* Have a history or presence of the signs and/or symptoms of urinary retention or benign prostatic hypertrophy.
* Show evidence of significant active neuropsychiatric disease or a history of suicidal thoughts or suicide attempt.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and sponsor's medical monitor.
* Have donated blood of more than 500 milliliters (mL) within 4 weeks prior to screening.
* Have an average weekly alcohol intake that exceeds 14 units per week or are unwilling to stop alcohol consumption 48 hours prior to check-in until the completion of the study (1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any participants unwilling to adhere to study caffeine restrictions.
* Have used any tobacco-containing or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to enrollment.
* Have consumed grapefruit or grapefruit-containing products 7 days prior to enrollment and during the study.
* Have a documented or suspected history of glaucoma.
* Participants determined to be unsuitable by the investigator for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2216684/Sertraline/LY2216684 + Sertraline: Period 1: LY2216684 18 milligram (mg) oral (po) dose on Days 1-3; Period 2: Sertraline 50 mg po dose on Day 4 followed by sertraline 100 mg po dose on Days 5-10; Period 3: LY2216684 18 mg po dose + sertraline 100 mg po dose on Days 11-13.
Period: Period 1: LY2216684 (Days 1-3)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 2
Period: Period 2: Sertraline (Day 4, 5-10)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Started | 18
Completed | 18
Not Completed | 0
Period: Period 3:LY2216684+Sertraline(Days11-13)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Started | 18
Completed | 17
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration-Time Curve Over a 24-Hour Dosing Interval (AUCτ) of LY2216684
Description: The Least Squares (LS) geometric mean AUCτ of LY2216684 was calculated based on the LY2216684 plasma concentration time curve from time 0 hour (hr) to time 24 hr (tau [τ]) when LY221684 was administered alone (Day 3) and when LY2216684 was coadministered with sertraline (Day 13). The Day 13-to-Day 3 ratio of the LY2216684 LS geometric mean of AUCτ and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 3 and Day 13
Population: The safety population included participants who were randomized, received study drug, and had at least 1 postdose safety assessment.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 18
hour*nanogram per milliliter (h*ng/mL)
  LY2216684 alone | 675 [618 to 738]
  LY2216684 + sertraline: number analyzed (Participants) | 13
  LY2216684 + sertraline | 792 [716 to 876]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.17, 90% CI 2-sided [1.06 to 1.30]

2. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of LY2216684
Description: The Least Squares (LS) geometric mean Cmax of LY2216684 was determined when LY2216684 was administered alone (Day 3) and when LY2216684 was coadministered with sertraline (Day 13). The Day 13-to-Day 3 ratio of the LY2216684 LS geometric mean of Cmax and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 3 and Day 13
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 18
nanogram per milliliter (ng/mL)
  LY2216684 alone | 65.9 [60.9 to 71.4]
  LY2216684 + sertraline: number analyzed (Participants) | 13
  LY2216684 + sertraline | 74.9 [68.1 to 82.4]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.14, 90% CI 2-sided [1.01 to 1.28]

3. Primary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Plasma Concentration (Tmax) of LY2216684
Description: Tmax of LY2216684 was determined using the median of paired differences between the 2 treatment groups when LY2216684 was administered alone (Day 3) and when LY2216684 was coadministered with sertraline (Day 13). The 90% confidence interval (CI) for the median of differences was calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 3 and Day 13
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 13
hours
  LY2216684 alone | 2.00 [2.00 to 4.00]
  LY2216684 + sertraline | 3.00 [2.00 to 4.00]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; p = 0.8281, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 1.00]

4. Primary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration-Time Curve Over a 24-Hour Dosing Interval (AUCτ) of Sertraline
Description: The Least Squares (LS) geometric mean AUCτ of sertraline was calculated based on the sertraline plasma concentration time curve from time 0 hour (hr) to time 24 hr (tau [τ]) when sertraline was administered alone (Day 10) and when sertraline was coadministered with LY2216684 (Day 13). The Day 13-to-Day 10 ratio of the sertraline LS geometric mean of AUCτ and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 10 and Day 13
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 17
hour*nanogram per milliliter (h*ng/mL)
  sertraline alone | 1240 [1090 to 1400]
  sertraline + LY2216684: number analyzed (Participants) | 13
  sertraline + LY2216684 | 1570 [1380 to 1790]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.27, 90% CI 2-sided [1.17 to 1.39]

5. Primary Outcome: Pharmacokinetic (PK) Parameter: Maximum Plasma Concentration (Cmax) of Sertraline
Description: The Least Squares (LS) geometric mean Cmax of sertraline was determined when sertraline was administered alone (Day 10) and when sertraline was coadministered with LY2216684 (Day 13). The Day 13-to-Day 10 ratio of the sertraline LS geometric mean of Cmax and the associated 90% confidence interval (CI) of the ratio were calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 10 and Day 13
Population: as for outcome 1
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 17
nanogram per milliliter (ng/mL)
  sertraline alone | 70.7 [62.4 to 80.1]
  sertraline + LY2216684: number analyzed (Participants) | 13
  sertraline + LY2216684 | 86.4 [75.6 to 98.7]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; ANOVA; Ratio of Geometric LS Means = 1.22, 90% CI 2-sided [1.10 to 1.36]

6. Primary Outcome: Pharmacokinetic (PK) Parameter: Time to Maximum Plasma Concentration (Tmax) of Sertraline
Description: Tmax of sertraline was determined using the median of paired differences between the 2 treatment groups when sertraline was administered alone (Day 10) and when sertraline was coadministered with LY2216684 (Day 13). The 90% confidence interval (CI) for the median of differences was calculated.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Day 10 and Day 13
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: hours
Arm/Group | LY2216684/Sertraline/LY2216684 + Sertraline
Number analyzed (Participants) | 13
hours
  sertraline alone | 6.00 [2.00 to 12.00]
  sertraline + LY2216684 | 8.00 [6.00 to 8.00]
Statistical Analysis 1: Comparison: LY2216684/Sertraline/LY2216684 + Sertraline; Test type: Superiority or Other; p = 0.3125, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 1.00, 90% CI 2-sided [0.00 to 2.00]

ADVERSE EVENTS:
Groups:
- LY2216684: Period 1: LY2216684 18 milligram (mg) oral (po) dose on Days 1-3; Period 2: Sertraline 50 mg po dose on Day 4 followed by sertraline 100 mg po dose on Days 5-10; Period 3: LY2216684 18 mg po dose + sertraline 100 mg po dose on Days 11-13.
- Sertraline: Period 2: Sertraline 50 mg po dose on Day 4 followed by sertraline 100 mg po dose on Days 5-10.
- LY2216684 + Sertraline: Period 3: LY2216684 18 mg po dose + sertraline 100 mg po dose on Days 11-13.
Arm/Group | LY2216684 | Sertraline | LY2216684 + Sertraline
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 11/20 | 6/18 | 13/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 (N=20) | Sertraline (N=18) | LY2216684 + Sertraline (N=18)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling of body temperature change (General disorders) | 6 (7) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Semenuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasodilatation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days